CLINICAL TRIAL: NCT07174310
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Intravenous Prasinezumab in Participants With Early-Stage Parkinson's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Intravenous (IV) Prasinezumab in Participants With Early-Stage Parkinson's Disease
Acronym: PARAISO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Prothena Biosciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BN44715; 2025-522683-32-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-12; First posted 2025-09-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prasinezumab (Experimental): Participants will receive Prasinezumab as an IV infusion in the double blind treatment period. Upon completion, eligible participants will enter into the Open Label Extension (OLE) phase.
  Interventions: Drug: Prasinezumab
- Placebo (Experimental): Participants will receive placebo as an IV Infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prasinezumab — Participants will receive Prasinezumab as an IV Infusion as per the schedule mentioned in the protocol.
  Arms: Prasinezumab
Drug: Placebo — Participants will receive Placebo as an IV Infusion per the schedule mentioned in the protocol
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics (PK) of prasinezumab compared with placebo in participants with early-stage Parkinson's disease (PD) on stable symptomatic monotherapy with levodopa.

ELIGIBILITY:
Inclusion Criteria:

* Body weight within 40-110 kilograms (kg) (88-242 pounds [lbs]) and a body mass index within the range 18-34 kg/m2
* Diagnosis of idiopathic PD based on Movement Disorder Society (MDS) criteria
* Has received monotherapy treatment
* An MDS-UPDRS Part IV score of 0 at screening and prior to randomization
* Hoehn and Yahr (H&Y) Stage 1 or 2 off medication at screening and prior to randomization
* Agreement to adhere to the contraception requirements

Exclusion Criteria:

* Pregnant or breastfeeding, or intention of becoming pregnant during the study or within the time frame in which contraception is required
* Medical history indicating a parkinsonian syndrome other than idiopathic PD
* Diagnosis of a significant neurologic disease other than PD
* Chronic uncontrolled hypertension

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to Confirmed Motor Progression Event on Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III Score | Up to at least Week 104

SECONDARY OUTCOMES:
Change From Baseline in Motor Function as Measured by the MDS-UPDRS Part III off Medication Score | Baseline, Week 104
Time to Worsening of Participants Motor Function as Reported by the Participant in the Presence of a Confirmed Motor Progression Event | Up to at least Week 104
Time to Meaningful Worsening in Clinician Global Impression of Change (CGI-C), Overall Disease Subscale | Up to at least Week 104
Time to increase in Levodopa Equivalent Daily Dose (LEDD) | Up to at least Week 104
Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) | From Baseline up to 70 days after the final study dose (up to at least Week 104)
Percentage of Participants With Adverse Events of Special Interest (AESI) | From Baseline up to 70 days after the final study dose (up to at least Week 104)
Percentage of Participants With Infusion Related Reactions (IRRs) | From Baseline up to 70 days after the final study dose (up to at least Week 104)
Percentage of Participants With Suicidal Ideation, as Measured by the Columbia-Suicide Severity Rating Scale (C-SSRS) | From Baseline up to 70 days after the final study dose (up to at least Week 104)
Serum Concentration of Prasinezumab | Predose and postdose at Baseline, Week 1, 4, 12, 24, 36, 52, 76, and after week 76 every 12 weeks thereafter until end of study (up to at least Week 104)
Percentage of Participants With Anti-drug Antibodies (ADAs) Against Prasinezumab at Baseline | At Baseline
Percentage of Participants With ADAs Against Prasinezumab During the Study | From Baseline up to 70 days after the final study dose (up to at least Week 104)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (19):
  - Neurology Center of North Orange County, Fullerton, California
  - Keck School of Medicine of USC, Los Angeles, California
  - Profound Research LLC at The Neurology Center of Southern California, Pasadena, California
  - UCSF Weill Institute for Neurosciences, San Francisco, California
  - Rocky Mountain Movement Disorders, Englewood, Colorado
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - JEM Research LLC, Atlantis, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - K2 - Villages, Lady Lake, Florida
  - K2 Medical Research-Maitland, Maitland, Florida
  - Charter Research - Winter Park/Orlando, Orlando, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Quest Research Institute, Farmington Hills, Michigan
  - Dent Neurological Institute, Amherst, New York
  - Weill Cornell Medical College, New York, New York
  - NeuroCare Center, Canton, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Central Texas Neurology Consultants, Round Rock, Texas
  - West Virginia University, Morgantown, West Virginia
- Canada (2):
  - CHUM, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- China (3):
  - West China Hospital of Sichuan University, Chengdu
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
  - The Second Affiliated Hospital of Suzhou University, Suzhou
- Poland (4):
  - NZOZ Vitamed, Bydgoszcz
  - Szpital Sw. Wojciecha, Gda?sk
  - Instytut Zdrowia Dr Boczarska-Jedynak Sp. z o.o. Sp. k., Oświęcim
  - NeuroProtect, Warsaw
- CNS - Campus Neurológico, Torres Vedras, Portugal
- Taiwan (2):
  - Changhua Christian Hospital, Changhua County
  - China Medical University Hospital, North Dist.
- United Kingdom (7):
  - Ninewells Hospital, Dundee- Scotland, Dundee
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Royal London Hospital, London
  - Charing Cross Hospital, London
  - Campus for Ageing and Vitality, Newcastle
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Plymouth Hospitals NHS Trust - Derriford Hospital, Plymouth,Devon

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing